CLINICAL TRIAL: NCT01062334
Title: Intraperitoneal Microdialysis Monitoring of Patients During the Early Postoperative Period After LAR With Reference to Early Diagnosis of Anastomotic Leakage Ore Other Complications
Brief Title: Peritoneal Microdialysis in Patients Undergoing Low Anterior Resection for Rectum Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Vejle Hospital (Other)
Responsible Party: Principal Investigator, Mark Ellebaek Pedersen, Doctor, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-20090147
Record Dates: First submitted 2010-01-28; First posted 2010-02-04 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Cancer
Keywords: Anastomotic leakage after LAR
MeSH Terms: conditions — Neoplasms

ARMS (1):
- Microdialysis (Experimental)
  Interventions: Procedure: Peritoneal Microdialysis, CT-scan, leakage scoring

INTERVENTIONS:
Procedure: Peritoneal Microdialysis, CT-scan, leakage scoring — Peritoneal microdialysis CT-scan before discharge Leakage scoring daily

SUMMARY:
Anastomotic leakage is a serious complication after LAR with high morbidity and mortality rates. Early diagnosis and treatment is mandatory. The primary aim of the present study is to investigate the clinical use of peritoneal microdialysis and whether is able to detect anastomotic leakage prior to clinical symptoms.

DETAILED DESCRIPTION:
Patients undergoing LAR for rectum cancer is subjected to peritoneal microdialyses during the postoperative period until the 7. postoperative day. Samples are collected every 4-hour. Samples will be analyzed continuously but the results will not be included in the clinical evaluation of the patient. Before removing the microdialysis catheter a CT whit rectal enema is preformed. Every day the patient will be evaluated whit a standardised clinical scoring system with attention at anastomotic leakage.

A total of 150 patients will be included in this study. The results of the peritoneal microdialyses will be compared with the clinical scorings system in each patient. The results form the uncomplicated courses will be used to define the normal variations in peritoneal microdialysis. This will be compared to results from patients with various complications.

The study is approved by the local scientific ethical committee No. ------

ELIGIBILITY:
Inclusion Criteria:

* Histological verified cancer
* The cancer must be located in rectum maximum of 15 cm.
* Diverting stoma is allowed
* Perioperative radio-chemotherapy is allowed

Exclusion Criteria:

* Disseminated cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-03; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Significant elevated peritoneal microdialysis parameter like lactate and L/P-ratio | Clinically complications with in 30th days after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Odense University hospital, Odense C, Fyn
  - Vejle hospital, Vejle